CLINICAL TRIAL: NCT03328403
Title: Endovascular Therapy in Acute Ischaemic Stroke Due to Large Vessel Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); Ruttonjee Hospital, Hong Kong (Unknown)
Responsible Party: Principal Investigator, Dr Anderson Chun-On Tsang, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 15-431
Record Dates: First submitted 2017-10-17; First posted 2017-11-01 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Acute Ischaemic Stroke
Keywords: Endovascular therapy; Mechanical thrombectomy; Acute ischaemic stroke treatment

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to use either the Aspiration System or one of the stent-retreivers (Trevo / Solitaire) first. Other devices would be used if the first device failed to open the occluded vessel satisfactorily, depending on clinical situation and the involved interventionists' preferences.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Aspiration First (Experimental): Aspiration thrombectomy with large bore catheters
  Interventions: Device: Aspiration First
- Stent retriever first (Experimental): Thrombectomy with a licensed stent retriever device
  Interventions: Device: Stent retriever first

INTERVENTIONS:
Device: Aspiration First — Use aspiration system (mainly Penumbra) first, other devices would be used if the first device failed to open the occluded vessel satisfactorily, depending on clinical situation and the involved interventionists' preferences.
  Arms: Aspiration First
Device: Stent retriever first — Use one of the stent retrievers (Trevo / Solitaire) first, other devices would be used if the first device failed to open the occluded vessel satisfactorily, depending on clinical situation and the involved interventionists' preferences.
  Arms: Stent retriever first

SUMMARY:
Aim of Study:

1. To develop a standardized patient selection criteria and imaging protocol for endovascular therapy in acute ischaemic stroke (AIS)
2. To create a local efficacy and safety database for intra-arterial mechanical thrombectomy devices use
3. To establish predictors for poor functional outcome despite successful recanalization

Study Design:

Prospective

Subject and Site:

100 acute ischaemic stroke patients with large vessel occlusion At Queen Mary and Ruttonjee Hospital, Hong Kong

Duration of participation:

2 years

Entry Criteria:

Subject must meet all inclusion criteria and none of the exclusion criteria

Consent:

Both English and Chinese versions of Informed consent are available and will be obtained from patient or his/her next of kin

DETAILED DESCRIPTION:
Our study aim to set a standard patient selection and imaging protocol based on previous positive trials for endovascular therapy in AIS patients. Local efficacy and safety data of the FDA mechanical devices mainly Penumbra Aspiration System and Solitaire Flow Restoration device will be collected to create a local database for future service development. Clinical predictors for poor clinical outcomes despite successful recanalization will be looked for.

Intra-arterial treatment consisted of arterial catheterization with a micro-catheter and micro-guide wire to the level of occlusion. Mechanical treatment could involve thrombus aspiration technique or use of a retrievable stent. The method of intra-arterial treatment will leave to the discretion of the involved interventionist. Only devices that have received U.S. Food and Drug Administration (FDA) or Conformite Europeenne (CE) approval will be used in the trial. One or more members of each intervention team have to have completed at least five full procedures with a particular type of device.

Outcome and Safety Measures:

The primary outcome is 90 days modified Rankin scale. The modified Rankin scale is a 7-point scale ranging from 0 (no symptoms) to 6 (death). A score of 2 or less indicates functional independence.

Secondary outcomes include:

1. NIHSS score at 24 hours and at 7 day or discharge if earlier
2. Activities of daily living measured using Barthel index and NIHSS at 90 days
3. Percentage of successful recanalization, defined as modified Thrombolysis in Cerebral Infarction (mTICI) of 2b (more that 50% of distal branches visible) or 3 (all distal branches visible) assessed at the end of procedure
4. Efficacy of work flow with time measure on onset to CT, CT to groin puncture, puncture to reperfusion and number of pass of device before successful recanalization
5. Final infarct volume measured by plain CT brain at 3 days after procedure
6. Death

ELIGIBILITY:
Inclusion Criteria:

* Onset: ≤ 4.5 hours from symptoms onset
* Age < 80
* Premorbid modified Rankin Score (mRS) ≤ 2
* NIHSS 8 - 29
* Clear and definite symptoms and signs suggesting stroke with hemiparesis as one of the presenting symptoms
* Plain CT brain showed no evidence of intracerebral haemorrhage and ASPECTS ≥ 7
* Multiphasic CT angiogram confirmed proximal vessel occlusion at internal carotid artery (ICA), carotid T junction, proximal middle cerebral artery (M1 segment to proximal M2 with loss of all M2 branches), proximal anterior cerebral artery (segment A1) or basilar artery

Exclusion Criteria:

* Interventionist or angio-laboratory not available
* Neurological signs rapidly resolving
* NIHSS>29
* Evidence of cerebral haemorrhage or subarachnoid haemorrhage on CT brain
* ASPECTS<7
* Excessive tortuosity of the vessel precluding device delivery
* Known chronic renal failure with creatinine level >250umol/L
* Known haemorrhagic diathesis
* Known coagulation factor deficiency
* Difficult blood pressure control with persistent systolic blood pressure >185mg or diastolic blood pressure >110mg despite aggressive blood pressure lowering therapy
* On anticoagulant and INR≥3
* On heparin in previous 48 hour and APTT>2x of normal
* Platelet counts <30
* Blood glucose <2.7mmol/L
* Known severe allergies to contrast medium
* Seizure as presenting symptoms with post-ictal hemiparesis
* Life expectancy < 3months
* Pregnant

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Modified Rankin scale | 90 days
  The primary outcome is 90 days modified Rankin scale. The modified Rankin scale is a 7-point scale ranging from 0 (no symptoms) to 6 (death). A score of 2 or less indicates functional independence.

SECONDARY OUTCOMES:
National Institute of Health Stroke Severity Score (NIHSS) | At 24 hours and at 7 day or discharge if earlier
  NIHSS score at 24 hours and at 7 day or discharge if earlier. NIHSS score describe the clinical severity of stroke symptoms, and is scored from 0 (no symptoms) to 42 (most severe deficits). The total NIHSS score before, at 24 hours after intervention and subsequent follow up will be assessed.
Activities of daily living | 90 days
  Activities of daily living measured using modified Barthel index (mBI). modified Barthel Index is a measurement of independence of daily living, the score ranges from 0 to 100, with higher score correlating to better outcome.
Percentage of successful recanalization | 1 day
  Percentage of successful recanalization, defined as modified Thrombolysis in Cerebral Infarction (mTICI) of 2b (more that 50% of distal branches visible) or 3 (all distal branches visible) assessed at the end of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mona Man-Yu Tse, MBBS, FHKAM, Principal Investigator — Queen Mary Hospital, Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong